CLINICAL TRIAL: NCT06370845
Title: Abundance of a Natural Odour in Human Cerebrospinal Fluid After Olfactory Exposure - the OLFO-Brain Study
Brief Title: Abundance of a Natural Odour in Human Cerebrospinal Fluid After Olfactory Exposure
Acronym: OLFO-Brain
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 0000-00000; kt24timper
Record Dates: First submitted 2024-03-21; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Overweight and Obesity
Keywords: natural odour Inhalation; RCT; Placebo Controlled; Cerebrospinal Fluid
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum (natural odour) (Active Comparator): Participants will inhale 50 uL of a natural odour contained in mini-inhaler over a period of 15 min.
  Interventions: Combination Product: Inhalation - Natural Odour
- Placebo Inhalation (Placebo Comparator): Participants will inhale 50 uL of placebo (propylene glycol) contained in mini-inhaler over a period of 15 min.
  Interventions: Combination Product: Inhalation - Placebo

INTERVENTIONS:
Combination Product: Inhalation - Natural Odour — Inhalation of 50 uL of a natural odour via nasal septum mini-inhaler.
  Arms: Verum (natural odour)
Combination Product: Inhalation - Placebo — Inhalation of 50 uL of Placebo via nasal septum mini-inhaler.
  Arms: Placebo Inhalation

SUMMARY:
The goal of this clinical trial is to investigate the abundance of a natural odour in human cerebrospinal fluid in obese and lean participants after inhalation thereof. Participants will undergo blood sample collection and inhalation of either a natural odour or placebo through an inhaler in addition to a liquor puncture prescribed in standard of care context.

ELIGIBILITY:
Inclusion Criteria Obese Participants:

* Age 18-60 years
* Written informed consent
* Scheduled for routine liquor puncture
* BMI ≥ 30 kg/m2
* No proven diagnose of diabetes

Inclusion Criteria Lean Participants:

* Age 18-60 years
* Written informed consent
* Scheduled for routine liquor puncture
* BMI 18-25 kg/m2

Exclusion Criteria:

* Known allergy to the natural odour
* Acute upper respiratory tract infection, acute or chronic sinusitis
* Present or past surgical intervention of the nasal cavity, the paranasal sinus, the pituitary or the frontal brain
* Pregnancy/lactation
* Any kind of severe chronic disease (e.g. severe heart failure, active cancer disease, severe renal impairment with an estimated glomerular filtration rate <30 ml/min/m2)
* Inability to understand the study procedure and to sign the study consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Detection of a natural odour in human CSF | 1 time assessment at baseline
  Detection of a natural odour in human CSF within 30 min following end of an 15 min olfactory stimulation thereof compared to placebo. The presence of the Verum (natural odour) will be assessed via Gas Chromatography-Mass Spectrometry. This will be analyzed using a binary logistic regression model to determine the odds ratio of detecting a natural odour in the CSF post-stimulation. The model will account for variables such as age, sex, and BMI category (obese vs. lean). The significance level will be set at p < 0.05.

SECONDARY OUTCOMES:
Abundance of a natural odour in human CSF of obese versus lean participants | 1 time assessment at baseline
  Detection of a natural odour in human CSF of obese versus lean participants within 30 min following end of an 15 min olfactory stimulation with a natural odour. Titration of the natural odour will be done via Gas Chromatography-Mass Spectrometry.
Change in abundance of a natural odour in blood before and after olfactory stimulation in relation to abundance in human CSF. | 2 times assessment at baseline (immediately before olfactory stimulation and within 30 min following end of olfactory stimulation)
  Change in abundance of a natural odour in blood before and after end (max 30 min) of an olfactory stimulation for 15 min in relation to abundance in human CSF. Titration of the natural odour in CSF and blood samples will be done via Gas Chromatography-Mass Spectrometry.
Change in abundance of a natural odour in blood before and after olfactory stimulation in obese as compared to lean participants. | 2 times assessment at baseline (immediately before olfactory stimulation and within 30 min following end of olfactory stimulation)
  Change in abundance of a natural odour in blood before and after end (max 30 min) of an olfactory stimulation for 15 min in obese as compared to lean participants. Titration of a natural odour in blood samples will be done via Gas Chromatography-Mass Spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Timper, Prof. Dr. med., Principal Investigator — University Hospital Basel, Department of Endocrinology, Diabetology and Metabolism
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Timper K, Bruning JC. Hypothalamic circuits regulating appetite and energy homeostasis: pathways to obesity. Dis Model Mech. 2017 Jun 1;10(6):679-689. doi: 10.1242/dmm.026609. PMID 28592656